CLINICAL TRIAL: NCT03817606
Title: A Comparison of Stryker's Tritanium Posterior Lumbar Cage and PEEK Implant on Spinal Fusion in Patients With Degenerative Disc Disease
Brief Title: A Comparison of Stryker's Tritanium Posterior Lumbar Cage and PEEK Implant
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to COVID-19 disruption
Sponsor: Riverside Medical Center (Other)
Collaborators: Stryker Spine (Industry)
Responsible Party: Principal Investigator, Juan Jimenez, Principal Investigator, Riverside Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RMC193
Record Dates: First submitted 2018-12-20; First posted 2019-01-25 (Actual); Results first posted 2021-12-15 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2022-12

CONDITIONS: Degenerative Disc Disease; Degenerative Scoliosis
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Intervention Model Description: Parallel randomized controlled trial
Who Masked: Participant
Masking Description: Study participants will not know which posterior lumbar cage they receive.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Tritanium Posterior Lumbar Cage (Experimental): Surgical placement of the Tritanium Posterior Lumbar Cage
  Interventions: Device: Tritanium Posterior Lumbar Cage
- AVS PEEK UniLIF (Active Comparator): Surgical placement of the AVS PEEK UniLIF Posterior Lumbar Cage
  Interventions: Device: AVS UniLIF PEEK Posterior Lumbar Cage

INTERVENTIONS:
Device: Tritanium Posterior Lumbar Cage — Placement of Tritanium Posterior Lumbar Cage via TLIF procedure
  Arms: Tritanium Posterior Lumbar Cage
Device: AVS UniLIF PEEK Posterior Lumbar Cage — Placement of AVS UniLIF PEEK Posterior Lumbar Cage via TLIF procedure.
  Arms: AVS PEEK UniLIF

SUMMARY:
The purpose of this study is to compare outcomes of patients with degenerative disc disease undergo lumbar spinal fusion with Stryker's Tritanium® Posterior Lumbar Cage or the UniLIF PEEK implant.

DETAILED DESCRIPTION:
This study protocol intends to examine the difference in efficacy between the Tritanium Posterior Lumbar Cage and the UniLIF PEEK implant with respect to how long it takes to achieve fusion of the spine. Study participants will undergo a transforaminal lumbar interbody fusion (TLIF) surgery and return for CT and x-ray follow-up to measure the degree to which fusion has been achieved. Survey methodology to assess perceived pain, level of disability, and quality of life will also be used to measure the differences between groups on these components.

ELIGIBILITY:
Inclusion Criteria:

* Subject is skeletally mature
* Subject has one or more of the following diagnoses:

  1. Degenerative Disc Disease (DDD) at one level or two contiguous levels from L2 to S1

     a. DDD may include up to Grade 1 spondylolisthesis at the involved level(s)
  2. Degenerative Scoliosis for which the interbody fusion device will be used as an adjunct to fusion
* Subject has received 6 months of non-operative therapy
* Subject understands the conditions of enrollment and is willing to sign and date the Informed Consent
* Subject agrees to comply with visit schedule and study assessments
* Provision of signed and dated informed consent form
* Subject stated willingness to comply with all study procedures and availability for the duration of the study
* Subject is in good general health as evidenced by medical history

Exclusion Criteria:

* Subject is obese (BMI > 40)
* Subject is sensitive to titanium materials
* Subject has an active infection at the operative site
* Subject has marked local inflammation
* Subject has any abnormality present which affects the normal process of bone remodeling including, but not limited to, severe osteoporosis involving the spine, bone absorption, osteopenia, tumors involving the spine, active infection at the site, or certain metabolic disorders affecting osteogenesis
* Subject has any mental, trauma, or neuromuscular disorder which would create an unacceptable risk of fixation failure or complications in postoperative care
* Subject has any open wounds
* Subject is pregnant or plans to become pregnant during the course of the study
* Subject has inadequate tissue coverage over the operative site.
* Subject has an neuromuscular deficit which places an unsafe load on the device during the healing period
* Subject has any condition of senility, mental illness, or substance abuse
* Subject has any other medical or surgical condition which would preclude the potential benefit of spinal implant surgery, such as the presence of tumors, congenital abnormalities, elevation of sedimentation rate unexplained by other diseases, elevation of white blood cell count (WBC), or marked left shift in the WBC differential count.
* Subject has prior fusion at the levels to be treated
* Subject is incarcerated

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2021-04-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Zipsie, Study Director — Riverside Medical Center; Juan Jimenez, MD, Principal Investigator — Riverside Medical Center
Locations (1):
- Riverside Medical Center, Kankakee, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tritanium Posterior Lumbar Cage | AVS PEEK UniLIF
Started | 2 | 2
Completed | 0 | 0
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- AVS PEEK UniLIF: Surgical placement of the AVS PEEK UniLIF Posterior Lumbar Cage
  AVS UniLIF PEEK Posterior Lumbar Cage: Placement of AVS UniLIF PEEK Posterior Lumbar Cage via TLIF procedure.
  Study not completed due to COVID-19
- Tritanium Posterior Lumbar Cage: Surgical placement of the Tritanium Posterior Lumbar Cage
  Tritanium Posterior Lumbar Cage: Placement of Tritanium Posterior Lumbar Cage via TLIF procedure
  Study not completed due to COVID-19.
- Total: Total of all reporting groups
Arm/Group | AVS PEEK UniLIF | Tritanium Posterior Lumbar Cage | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Continuous [Mean (Full Range); unit: years] | 64 [61 to 67] | 53.5 [53 to 54] | 58.75 [53 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants] — Data collection was not completed as the study did not progress due to COVID-19 Population: The patients were enrolled; however, the study was not completed. No participants completed the study. There was no data to analyze.
  Participants
    United States | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Fusion Success
Description: CT and X-ray imaging will be obtained at study visits and Fusion Success will be defined by the following criteria: no lucent area around the implant; no presences of herniated disk, central stenosis, lateral recess stenosis, foraminal stenosis, facet anthropathy; no fracture of the device, graft or vertebra; visible bone formation in or about the graft material; less than 3 degrees of inter-segmental position change on flexion and extension views; presence of subsidence: a migration of more than 3mm into the adjacent vertebra; and the proportion of bridging bone visually estimated over the surface area of the joint
Time Frame: 12 Months
Population: Four patients were initially enrolled; however, due to COVID-19, study enrollment was suspended and patient follow up was limited to standard of care. The study was not continued. No data to analyze.
Arm/Group | AVS PEEK UniLIF | Tritanium Posterior Lumbar Cage
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Change in Visual Analogue Scale
Description: Change in low back pain as indicated by Visual Analogue Scale (VAS). The VAS measures subjects' self-reported pain level on a 100 mm line on which the subject indicates their level of pain, where 0 is no pain and 100 is worst imaginable pain.
Time Frame: Baseline; 6 weeks; 3 months; 6 months; and 12 months post operation
Population: Four patients were initially enrolled; however due to COVID-19 enrollment was suspended and patient follow up was limited to standard of care. The study was not continued. No Data to Analyze
Arm/Group | AVS PEEK UniLIF | Tritanium Posterior Lumbar Cage
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change in Low Back Function
Description: Change in Oswestry Disability Index (ODI) score. The ODI assesses disability related to lower back pain using a Likert 0 to 5 scale. There are 10 sections to the assessment, and the scores are represented as a percentage ranging from 0 (no disability) to 100 (completely disabled).
Time Frame: Baseline; 6 weeks; 3 months; 6 months; and 12 months post operation
Population: as for outcome 2
Arm/Group | Tritanium Posterior Lumbar Cage | AVS PEEK UniLIF
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change in Quality of Life: SF-36 PCS
Description: Change in perception of quality of life, as measured by Short Form 36 Health Survey (SF-36 PCS). The SF-36 PCS is a 36-item patient reported health questionnaire to measure perceived quality of life across 8 domains. Higher scores indicate higher quality of life, and lower scores indicate lower quality of life. Scores range from 5 (poor physical function) to 80 (excellent clinical function).
Time Frame: Baseline; 6 weeks; 3 months; 6 months; and 12 months post operation.
Population: as for outcome 2
Arm/Group | Tritanium Posterior Lumbar Cage | AVS PEEK UniLIF
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Number of Participants That Return to Work
Description: Subjects who were unable to work due to their back pain who return to work.
Time Frame: Baseline; 6 weeks; 3 months; 6 months; and 12 months post operation
Population: as for outcome 2
Arm/Group | Tritanium Posterior Lumbar Cage | AVS PEEK UniLIF
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Ambulatory Status
Description: Amount of time to full ambulation without assistance for study participants who had no or partial ambulation at baseline.
Time Frame: Baseline; 6 weeks; 3 months; 6 months; and 12 months post operation
Population: as for outcome 2
Arm/Group | Tritanium Posterior Lumbar Cage | AVS PEEK UniLIF
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Number of Participants With Serious Adverse Events
Description: Any event meeting the Serious Adverse Event reporting criteria detailed in the study protocol occurring at the following time intervals: TLIF procedure, hospital recovery and discharge, and 6 weeks-, 3 months-, 6 months- and 12 months post operation
Time Frame: 6 weeks; 3 months; 6 months; and 12 months post operation
Population: as for outcome 2
Arm/Group | Tritanium Posterior Lumbar Cage | AVS PEEK UniLIF
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Change in Quality of Life: EQ-5d
Description: Change in perception of quality of life, as measured by the EuroQol-5d (EQ-5d). The EuroQol-5d is a five question broad quality of life measure that can be combined into a single index and represents current health. A score of 0.0 is the worst imaginable health while a score of 1.0 would be the best imaginable health.
Time Frame: Baseline; 6 weeks; 3 months; 6 months; and 12 months post operation
Population: as for outcome 2
Arm/Group | Tritanium Posterior Lumbar Cage | AVS PEEK UniLIF
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Tritanium Posterior Lumbar Cage | AVS PEEK UniLIF
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 0/2 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-09-21): https://cdn.clinicaltrials.gov/large-docs/06/NCT03817606/Prot_000.pdf
  • Informed Consent Form (2018-10-08): https://cdn.clinicaltrials.gov/large-docs/06/NCT03817606/ICF_001.pdf